CLINICAL TRIAL: NCT02699008
Title: High On-treatment Platelet Reactivity to Adenosine Diphosphate Identified by Multiple Platelet Function Assay Guide to Modify Anti-platelet Strategy in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: High On-treatment Platelet Reactivity Identified by Multiple Platelet Function Assay
Acronym: HOPEmultiPFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFT-2015-01
Record Dates: First submitted 2015-10-30; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Acute Coronary Syndrome
Keywords: clopidogrel；antiplatelet therapy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HPR-Ticagrelor row (Active Comparator): ACS patients aftergoing PCI treated with clopidogrel and aspirin were included. in the 3-5th day after prescription of clopidogrel, platelet function were tested simultaneously by three methods: Light transmittance aggregometry（LTA）, Thrombelastography (TEG) ,Innovance PFA-200 . According to three method results（Two of three or all three results higher than cutoff value was identified as HPR, MPALTA>50%;MAADP>47mm;CTP2Y<106s）.Patients was defined as HPR and unHPR, HPR patients were randomized divided into HPR-Ticagrelor(HPR-T) and HPR-Clopidogrel(HPR-C)
  Interventions: Drug: Ticagrelor
- HPR-Clopidogrel row (Active Comparator): Thrombelastography (TEG) ,Innovance PFA-200 . According to three method results（Two of three or all three results higher than cutoff value was identified as HPR, MPALTA>50%;MAADP>47mm;CTP2Y<106s）.Patients was defined as HPR and unHPR, HPR patients were randomized divided into HPR-Ticagrelor(HPR-T) and HPR-Clopidogrel(HPR-C)
  Interventions: Drug: Clopidogrel
- unHPR row (Active Comparator): Thrombelastography (TEG) ,Innovance PFA-200 . According to three method results（Two of three or all three results higher than cutoff value was identified as HPR, MPALTA>50%;MAADP>47mm;CTP2Y<106s）.Patients was defined as HPR and unHPR, HPR patients were randomized divided into HPR-Ticagrelor(HPR-T) and HPR-Clopidogrel(HPR-C)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Antiplatelet agent
  Arms: HPR-Clopidogrel row; unHPR row
Drug: Ticagrelor — New P2Y12 receptor inhibitor antiplatelet agent
  Arms: HPR-Ticagrelor row

SUMMARY:
High on-treatment platelet reactivity to adenosine diphosphate was a important reason to cause ischemic events in antiplatelet therapy. Using single testing to definite HPR may miss the "true HPR" or over estimate HPR, which may lead to randomized trials failed. It is not known whether combined multiple platelet function testing could assist to ensure"ture"HPR and improve clinical outcomes.

DETAILED DESCRIPTION:
This was a single-center, randomized, prospective study. ACS patients undergoing PCI treated with clopidogrel and aspirin were included. in the 3-5th day after prescription of clopidogrel, platelet function were tested simultaneously by three methods: MPAADP by Light transmittance aggregometry（LTA）, MAADP by Thrombelastography (TEG) ,and CTP2Y by Innovance PFA-200 . According to three result（Two of three or all three results higher than cutoff value was identified as HPR, MPALTA>50%;MAADP>47mm;CTP2Y<106s）.Patients was defined as HPR(n=125) or unHPR(n=232), HPR patients were divided into HPR-Ticagrelor(HPR-T)and HPR-Clopidogrel(HPR-C) randomized. HPR-T group(n=77) patients' antiplatelet agents changed to ticagrelor, both unHPR and HPR-C groups keep unchanged(Clopidogrel). The major adverse cardiovascular events (MACE) were recorded during 1 year Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ACS patients（UAP;USTEMI,STEMI）
* Undergoing PCI
* Oral antiplatelet therapy

Exclusion Criteria:

* Stable CAD

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 1 year
  stent thrombosis；ACS；all cause Death；stroke；

SECONDARY OUTCOMES:
Bleeding events | 1 year
  gastrointestinal bleeding；gastrointestinal bleeding；other bleeding need RBC transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Zhou xin, MD, Study Chair — Wuhan Asia Heart Hospital
Locations (1):
- Wuhan Asia Heart Hospital, Wuhan, Hubei, China